CLINICAL TRIAL: NCT05072249
Title: A Multi-national, Prospective Mixed Methods Study of the Effectiveness of Naloxone (Including Intranasal Nyxoid) Administration by Lay People in Reversing Opioid Overdose
Brief Title: European Cohort Study of the Effectiveness of Take Home Naloxone
Acronym: NalPORS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: MR903 9501
Record Dates: First submitted 2021-06-08; First posted 2021-10-08 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Opioid Overdose
Keywords: overdose; take home naloxone; opioids; effectiveness; prevention; fatalities; mixed methods
MeSH Terms: conditions — Opiate Overdose; Drug Overdose; Death | interventions — Naloxone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lay person provided with take home naloxone: Naloxone all forms
  Interventions: Drug: Naloxone

INTERVENTIONS:
Drug: Naloxone — Take Home Naloxone for reversing opioid overdose
  Other Names: Prenoxad; Nyxoid; Ventizolve

SUMMARY:
This study aims to assess the effectiveness of take-home naloxone (THN) to reverse opioid overdose when administered by lay persons in a real world setting. This multicentre, prospective, observational cohort study will be conducted across Europe using a mixed method approach. Recruiting 6000 individuals to whom a supply of THN has been provided, for n=600 to witness an opioid overdose. The co-primary outcomes are to determine the rate of administration of naloxone and frequency of deaths in the 24 hours subsequent to the administration of naloxone. This will be captured through structured interviews with those who report witnessing an opioid overdose in the 6 month study period, approximately n=600, to elicit further information on the overdose and any naloxone administered. Naloxone training materials and education provided will be examined through questions in the structured interview. In-depth qualitative interviews will also be conducted with 60 participants who have witnessed an overdose, in order to better understand the use, safety and effectiveness of different naloxone products (particularly Nyxoid). As part of the qualitative analysis, interview transcripts will be assessed by an expert clinician panel for accuracy of diagnosis, actions taken and aftercare. Routine data from national health registers will be used to gather mortality data. This study will report on the use of different formulations of naloxone. In addition, this study serves as a Post Authorisation Efficacy Study (PAES) for the intranasal (IN) naloxone, Nyxoid developed by MundiPharma and focuses on drug safety and training.

DETAILED DESCRIPTION:
Accidental opioid overdose is a global crisis. Naloxone is an accessible, safe and effective antidote for this preventable cause of mortality. While it has been used to treat opioid overdose in hospital and pre-hospital settings since the 1970s, take home naloxone programmes have been introduced more recently after opioid users were recognised as potential first responders. This study aims to assess the effectiveness of take-home naloxone (THN) to reverse opioid overdose when administered by lay persons in a real world setting. This multicentre, prospective, observational cohort study will be conducted across Europe using a mixed method approach, recruiting 6000 individuals to whom a supply of THN has been provided (comprising four groups:1. patients in treatment for opioid use disorder (OUD), 2. Individuals using opioids but out-of-treatment, 3. family members, friends and other close carers, and 4. staff working with individuals with OUD) for n=600 to witness an opioid overdose. The co-primary outcomes are to determine the rate of administration of naloxone and frequency of deaths in the 24 hours subsequent to the administration of naloxone.

This will be captured through two stages and two sub-studies. Main study stage 1: All consenting participants (n=6,000) will be asked to complete an enrolment questionnaire with the member of staff recruiting them into the study. In addition, the staff member will be asked to complete a brief record of the naloxone and training provided to the participant. Participants will be texted monthly to prompt them to contact research staff if they have witnessed an opioid overdose. Staff who have frequent or regular contact with participants (including instances when a replenishment of naloxone is given) will also prompt participants to make contact with research staff to notify them of a witnessed opioid overdose. All participants will be contacted at six months and asked to take part in a structured interview. In addition, national/regional death registers will be probed to confirm mortality data for study participants who are at risk of experiencing an opioid overdose themselves.

Main study, Stage 2: Participants who report that they have witnessed an opioid overdose during the six-month follow-up period will be asked to take part in a structured interview with a researcher about this witnessed overdose to capture our primary outcomes (approximately n=600).

Sub-study A: comprises two structured surveys incorporated into a) the Enrolment training information form (to examine naloxone training and materials provided) and b) the Stage 2 Interview completed by participants who have witnessed an overdose (to ask about the extent they followed the nasal naloxone Nyxoid Quick Start Guide (QSG) (or equivalent instructions). The questions are designed to better understand the effectiveness of the Nyxoid nasal naloxone educational and training materials delivered to participants who were provided with Nyxoid nasal naloxone and who were subsequently present at an overdose.

Sub-study B: comprises qualitative interviews with 60 UK participants who witness a diverse range of overdose events of the approx. n=600 (Main Study Stage 2). The aim of sub-study B is to better understand the use, safety, and effectiveness of different naloxone products. Qualitative interviews will be guided by a topic guide and conducted by telephone. The topic guide will capture details of any overdoses experienced or witnessed since the study started before focusing in more depth on the most recent overdose witnessed. Participants will also be asked about any training they have had, or need, in naloxone administration. In addition, a clinical expert assessment of the accurate identification of an opioid overdose and the participant's response to the opioid overdose (as detailed in the transcribed interviews) will be performed and documented. Answers will be assessed by an expert clinician panel for accuracy of diagnosis, actions taken and aftercare.

This study will report on the use of different formulations of naloxone, and different national systems of training and provision. In addition, this study serves as a Post Authorisation Efficacy Study (PAES) for the intranasal (IN) naloxone, Nyxoid developed by Mundipharma and focuses on drug safety and training.

ELIGIBILITY:
Inclusion Criteria:

* Member of at least one of the groups above (a-d)
* Aged ≥18 years
* Provided with THN supply at time of enrolment (or can demonstrate that they have a supply of THN (in-date) and have received training at time of enrolment).
* Have access to reliable mobile telephone and can present it.
* Willing to participate in follow-up
* Who have provided written informed consent.

Exclusion Criteria:

The following persons will be excluded:

* Needs an interpreter
* Already entered the study
* Not willing or able to partake in follow-up telephone survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any of below:
  1. Patients in treatment for opioid use disorder (OUD)
  2. Out-of-treatment individuals with OUD
  3. Family members, friends and other close carers of individuals with OUD
  4. Staff working with individuals with OUD
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of deaths in the 24 hours or later if information is available subsequent to administration of naloxone by lay-persons to reverse an opioid overdose in the real world. | Ongoing - over six months period post enrolment (at most recent overdose witnessed)
  frequency of deaths among those witnessing opioid overdose (n=600)
Administration rate of THN with the intention of reversing an opioid overdose by lay persons provided with THN who witness an opioid overdose. | Ongoing -over six months period post enrolment (at most recent overdose witnessed)
  Rate of THN administration among those witnessing opioid overdose (n=600)

SECONDARY OUTCOMES:
Percentage of participants who indicate carrying THN (on day of interview) | Ongoing over 6-month period post enrolment
  Percentage (n=6000)
Percentage of participants who witness an opioid overdose over 6-month period. | Ongoing over 6-month period post enrolment
  Percentage (n=6000)
Confirm death or survival of participants | On-going over 6 month period post enrolment
  percentage (n=600)
Percentage of participants who witness an opioid overdose who report there was THN present | Ongoing over 6-month period post enrolment (at most recent overdose witnessed)
  Percentage (n=600)
Percentage of participants who are carrying THN when witness an opioid overdose | Ongoing over 6-month period post enrolment (at most recent overdose witnessed)
  Percentage (n=600)
Percentage of participants who witness an opioid overdose, where there was THN present, and administer THN | Ongoing over 6-month period post enrolment (at most recent overdose witnessed)
  Percentage (n=600)
Percentage of participants who witness an overdose and administer THN who report respiratory depression occurred in person they resuscitated within one hour of administering THN | On-going within 6-month period post enrolment (at most recent overdose witnessed)
  Percentage (n=600)
Percentage of participants who witness an overdose, who report a second dose of naloxone administered to a person experiencing an opioid overdose within 1-hour post administration of first dose of THN | 6-month follow-up (at most recent overdose witnessed)
  Percentage (n=600)
Percentage of participants who report withdrawal symptoms (including anger, rage and violence) occurred in person they resuscitated with THN | On-going over 6-month period post enrolment (at most recent overdose witnessed)
  Frequency of each symptom witnessed (n=600) (at most recent overdose witnessed)
Percentage of participants witnessing an overdose where the person receiving naloxone has survived at 2 hours post administration of naloxone OR at arrival of ambulance/medical assistance if this occurs before 2 hours have passed since opioid overdose | Ongoing over 6-month period post enrolment
  Percentage (n=600)
Percentage of participants who witness an opioid overdose and report fatal outcomes within 2 hours of identification of opioid overdose or at arrival of ambulance/medical assistance a) of witnessed opioid overdoses b) Of witnessed opioid overdoses | Ongoing over 6-month period post enrolment
  Percentage (n=600)
Percentage of participants who witness an overdose who correctly diagnosed opioid overdose crisis-through multiple response questions | Ongoing interviews 6-month post enrolment follow-up
  Percentage (n=600)
Percentage of participants who witness an opioid overdose who correctly diagnose opioid overdose crisis-through multiple response questions | Ongoing interviews 6-month post enrolment follow-up
  Percentage (n=600)
Percentage of participants who witness an opioid overdose who correctly respond to opioid overdose crisis-through multiple response questions | Ongoing interviews 6-month post enrolment follow-up
  Percentage (n=600)

OTHER OUTCOMES:
Percentage of participants that received various forms of Nyxoid training materials during their naloxone training (patient information card, training video, information on leaflet and images in nyxoid pack). | Enrolment & Stage 1 interview conducted at 6 months
  Percentage (n=3000 (only those receiving nyxoid))
Percentage of participants (receiving nyxoid) that appropriately recognised and responded to an overdose. | Ongoing interviews 6-months post enrolment follow-up
  Percentage (n=300 (only those receiving nyxoid witnessing O/D)
Percentage of participants (receiving nyxoid) that appropriately responded to an overdose. | Ongoing interviews 6-months post enrolment follow-up
  percentage (n=300)
Percentage of participants that had received nyxoid naloxone training prior to enrolling | Enrolment
  Percentage (n=3000)
Positive response given (by those receiving nyxoid) stating no improvement after 2-3 minutes OR overdose symptoms come back | Ongoing interviews 6-months post enrolment follow-up
  Percentage (n=300)
Percentage of participants (receiving nyxoid) that inappropriately responded to an overdose. | Ongoing interviews 6-months post enrolment follow-up
  Percentage (n=300)
Increased understanding of carriage of naloxone products and disposal of used kits | 6-month follow-up (at most recent overdose witnessed)
  Qualitative interview with those having witnessed an opioid overdose from UK n=60
Increased understanding of how naloxone is administered in an emergency overdose situation, including any problems encountered (e.g. device malfunction or misuse) | 6-month follow-up (at most recent overdose witnessed)
  Qualitative interview with those having witnessed an opioid overdose from UK n=60
Increased understanding of decision making processes relating to naloxone administration in an emergency opioid overdose situation, including giving/not giving a second dose | 6-month follow-up (at most recent overdose witnessed)
  Qualitative interview with those having witnessed an opioid overdose from UK
Increased understanding of the impact of the social and environmental setting in which the overdose occurs - on naloxone use | 6-month follow-up (at most recent overdose witnessed)
  n=60 qualitative interview with those having witnessed an opioid overdose from UK n=60
Increased understanding of the links between naloxone carriage and use on willingness to call an ambulance when witnessing an opioid overdose | 6-month follow-up (at most recent overdose witnessed)
  Qualitative interview with those having witnessed an opioid overdose from UK n=60
Increased understanding of the effectiveness of naloxone administration, including speed of reversal and opioid overdose outcome | 6-month follow-up (at most recent overdose witnessed)
  Qualitative interview with those having witnessed an opioid overdose from UK n=60
Increased understanding of any negative consequences of naloxone administration (e.g. victim withdrawals, aggression, respiratory depression and death) and their implications for future opioid overdose events witnessed | 6-month follow-up (at most recent overdose witnessed)
  Qualitative interview with those having witnessed an opioid overdose from UK n=60
Increased understanding of care of the victim both during the opioid overdose and post-naloxone administration | 6-month follow-up (at most recent overdose witnessed)
  Qualitative interview with those having witnessed an opioid overdose from UK n=60
Increased understanding of knowledge of naloxone, including training and information needs | 6-month follow-up (at most recent overdose witnessed)
  Qualitative interview with those having witnessed an opioid overdose from UK n=60
Increased understanding of views on the THN training materials | 6-month follow-up (at most recent overdose witnessed)
  Qualitative interview with those having witnessed an opioid overdose from UK n=60
Accurate diagnosis of Opioid overdose. | 6-month follow-up (at most recent overdose witnessed)
  Expert assessment of transcripts of qualitative interviews using non-validated naloxone administration scale. 5-point Likert scale (1 (very low)- 5 (very high)
Accurate identification of respiratory depression. | 6-month follow-up (at most recent overdose witnessed)
  Expert assessment of transcripts of qualitative interviews using non-validated naloxone administration scale. 5-point Likert scale (1 (very low)- 5 (very high).
Appropriate response to opioid overdose | 6-month follow-up (at most recent overdose witnessed)
  Expert assessment of transcripts of qualitative interviews using non-validated naloxone administration scale. 5-point Likert scale (1 (very low)- 5 (very high)
Adequate post naloxone aftercare. | 6-month follow-up (at most recent overdose witnessed)
  Expert assessment of transcripts of qualitative interviews using non-validated naloxone administration scale. 5-point Likert scale (1 (very low)- 5 (very high)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Sir John Strang, Principal Investigator — King's College London
Locations (6):
- SundhedsTeam, Socialforvaltningen, Københavns Kommune, Copenhagen, Denmark
- Stockholm Centre for Dependency Disorders, Stockholm, Sweden
- United Kingdom (4):
  - Birmingham and Solihull Mental Health Foundation Trust, Birmingham
  - Public Health Wales, Cardiff
  - Scottish Drugs Forum, Glasgow
  - South London and the Maudsley, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metrebian N, Carter B, Eide D, McDonald R, Neale J, Parkin S, Dascal T, Mackie C, Day E, Guterstam J, Horsburgh K, Kaberg M, Kelleher M, Smith J, Thiesen H, Strang J. A study protocol for a European, mixed methods, prospective, cohort study of the effectiveness of naloxone administration by community members, in reversing opioid overdose: NalPORS. BMC Public Health. 2023 Aug 24;23(1):1608. doi: 10.1186/s12889-023-16445-6. PMID 37612698